CLINICAL TRIAL: NCT03999541
Title: Fresh Versus Frozen Embryos for Infertility in the Poor Responders as Defined by the Bologna Criteria
Brief Title: Freeze-all Policy in Poor Responders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Al-Yasmeen Fertility and Gynecology Center (Other)
Responsible Party: Principal Investigator, Yasmin Magdi, Director, Al-Yasmeen Fertility and Gynecology Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: #0014
Record Dates: First submitted 2019-06-22; First posted 2019-06-26 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Masking Description: Blinding of the allocated intervention is not possible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Freeze-all (Experimental): Good quality embryos (either day 3 or 5) will be frozen and subsequent frozen embryo transfer will be arranged within three months of the egg retrival.
  Interventions: Other: Freeze-all policy
- Fresh embryo transfer (No Intervention): Women will undergo fresh embryo transfer at the cleavage (day 3) or blastocyst stage (day 5).

INTERVENTIONS:
Other: Freeze-all policy — A policy of freezing all the embryos followed by subsequent thawed frozen embryo transfer
  Arms: Freeze-all

SUMMARY:
To compare the effects of fresh embryo transfers (ET) and elective frozen-thawed embryo transfer cycles in poor ovarian responders.

ELIGIBILITY:
Inclusion Criteria:

* All patients that fulfill the Bologna criteria [at least 2 of the following 3 features must be present: (i) advanced maternal age or any other risk factor for POR; (ii) a previous POR; and (iii) an abnormal ovarian reserve test (ORT)]
* if the progesterone serum level was ≤1.5 ng/mL on the trigger day.
* body mass index 18-32 kg/m2
* Both partners are able to provide written informed consent.
* At least 1 good quality embryo on day 3 after egg collection on day 3 according to the Istanbul consensus (7-8 cells; with symmetric blastomeres and <10% fragmentation by volume).
* Endometrial thickness ≥8 mm on trigger day.
* a normal uterine cavity on ultrasound.
* IVF/ICSI with only fresh semen

Exclusion Criteria:

* Pre-implantation genetic testing is being planned.
* if they had severe endometriosis, uterine pathology (myomas, adenomyosis, endocrinopathies, adhesions, acquired or congenital abnormalities), untreated tubal hydrosalpinges, ovarian tumor, recurrent spontaneous abortion, implantation failure after ≥ 2 fresh or frozen ET.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 178 (Estimated)
Dates: Start 2019-07-30 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Livebirth rate | 32 weeks
  The proportion of women in the population who had at least one live baby.

SECONDARY OUTCOMES:
Pregnancy rate | 2 weeks
  Positive pregnancy test at two weeks +/- three days after embryo transfer
Clinical pregnancy rate | 6-8 weeks
  The presence of at least one fetal heartbeat at ultrasound between six and eight weeks of gestation

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Yasmeen Fertility and Gynecology Center, Banhā, Egypt

IPD SHARING:
Plan to Share IPD: Yes